CLINICAL TRIAL: NCT01227980
Title: Corticotropin-Releasing Hormone Receptor 1 (CRH1) Antagonism in Anxious Alcoholics
Brief Title: Corticotropin-Releasing Hormone Receptor 1 (CRH1) Antagonism in Anxious Alcoholics^
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110010; 11-AA-0010 (Other: NIH)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Alcohol-Related Disorders; Alcohol Dependence; Alcoholism; Anxiety Disorder
Keywords: Addiction; Alcohol; Alcohol Treatment; Alcoholics; Alcohol Dependence; Anxiety Disorder; Alcoholism
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Anxiety Disorders; Behavior, Addictive | interventions — pexacerfont

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pexacerfont (Active Comparator): Pexacerfont was given orally as a loading dose of 300 mg/day for 1 week, followed by 100mg/day for 16-20 days
  Interventions: Drug: Pexacerfont
- Placebo (Placebo Comparator): Oral placebo was given during the 1-week loading dose phase, and during the next 16-20 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pexacerfont — 300 mg, orally, once/day during week 1, 100 mg, orally, once/day during weeks 2 and 3.
  Arms: Pexacerfont
Drug: Placebo — 300 mg, orally, once/day during week 1, 100 mg, orally, once/day during weeks 2 and 3.
  Arms: Placebo

SUMMARY:
Background:

- Individuals who are dependent on alcohol often have feelings of anxiety, irritability, anger, and depression. These feelings, as well as stress, may contribute to the risk of relapse and continued drinking. Studies have shown that alcohol consumption increases the activity of certain molecules in the brain known as CRH1 receptors, which are key to producing the body s response to stress, and whose activation generates feelings of anxiety. Researchers are interested in learning whether the experimental drug pexacerfont, which blocks CRH1 receptors and has been studied in individuals with anxiety disorders and depression, can lessen anxiety and craving for alcohol as part of alcohol-dependence treatment.

Objectives:

- To determine the safety and effectiveness of pexacerfont as a treatment for anxiety-related alcohol craving.

Eligibility:

- Individuals between 21 and 65 years of age who are alcohol-dependent and have problems with anxiety.

Design:

* This study requires an inpatient admission to the NIH Clinical Center for approximately 1 month, with two additional study visits 1 week and 1 month after discharge from the hospital.
* Participants will be screened with a medical history, physical examination, and blood and urine tests.
* During the inpatient period, participants will have standard treatment for alcohol dependence, including support and interventions from institute staff to address cravings, anxiety, or other psychological problems. Participants will not receive formal psychological treatment or psychiatric medications for anxiety, but will receive training in relaxation techniques.
* Participants will be assigned to take either pexacerfont or placebo for 3 weeks. During this time, participants will have the following procedures:
* Frequent blood tests.
* Rating scales and questionnaires about alcohol cravings and anxiety.
* Dexamethasone suppression test with frequent blood draws to study hormone response to stress.
* Social stress test involving public speaking, followed by blood samples and questionnaires on alcohol craving.
* Cue Reactivity (CR) session to study cravings and responses to alcohol-based cues.
* Functional magnetic resonance imaging scan to evaluate brain activity while taking the medication or placebo.
* Participants will have two follow-up visits for additional blood tests and questionnaires about the effects of the treatment ^.

DETAILED DESCRIPTION:
OBJECTIVE :

To evaluate pexacerfont, an orally available, brain penetrant selective CRH1 antagonist for its ability to modulate emotional and motivational processes in anxious, recently detoxified alcohol dependent patients.

STUDY POPULATION:

Up to 70 anxious, alcohol dependent subjects, aged 21-65 years will be enrolled to complete the study in 50 patients.

DESIGN

Subjects will be inpatients and enter the present protocol once withdrawal treatment, if needed, is completed. They will undergo interviews for construction of guided imagery scripts during a 3 day pre-treatment phase, after which they will receive randomized double blind treatment with active medication or placebo for 23 days, followed by a 3 day post-treatment inpatient monitoring phase, and two follow-up outpatient visits. While hospitalized, repeated measures of spontaneous craving for alcohol, ratings of psychopathology, and blood chemistry including cortisol will be obtained over this time. During the second week of treatment, craving responses will be assessed in a challenge session that combines a social stressor and exposure to physical alcohol cues. During the final week, three sessions of guided imagery will be carried out, on separate days and in a counter-balanced order, exposing the subject to personalized stress-, alcohol- or neutral condition associated stimuli. The final week will also include an fMRI session with emotional and motivational tasks, on a day separate from any guided imagery session. Subjects will remain hospitalized throughout the study, will remain on the unit for a 3 day post-medication monitoring period, and will return for follow up app. 1 and 4 weeks following completion of randomized treatment.

OUTCOME MEASURES

The primary outcome will be craving for alcohol on guided imagery challenge sessions. Secondary outcomes will include craving as measured in the combined social stress alcohol cue challenge session, spontaneous craving and psychopathology ratings repeatedly measured on the inpatient unit over time. Exploratory blood biomarkers and brain responses to positive and negative affective stimuli on the fMRI session will also be obtained.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Signed written informed consent:

     a. Patients must be competent to understand the nature of the study, sign the informed consent prior to any study-related procedures, agree to comply with the prescribed dosage regimens, agree to remain hospitalized at the NIH Clinical Center throughout the duration of the study and to return for follow-up visits as specified, and agree to communicate to study personnel about adverse events and concomitant medication use.
  2. Target population:

     1. DSM-IV diagnosis of alcohol dependence on SCID interview,
     2. alcohol problems as primary complaint among substance use disorders,
     3. alcohol use within the last month.
     4. Spielberger trait anxiety inventory score > 39.
     5. Right-handedness
  3. Age and sex:

     1. Men and women, ages 21 65 years.
     2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) prior to enrollment, and agree to using an adequate method of contraception to avoid pregnancy for a period of 6 months beginning from first dose of randomized treatment. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Adequate methods of contraception are practicing complete abstinence from intercourse for two weeks prior to administration of study drug; having a male sexual partner(s) who is surgically sterilized (vasectomy with documentation of azoospermia) prior to inclusion; having a sexual partner(s) who is/are exclusively female; using oral contraceptives (either combined or progestogen only) with single-barrier method of contraception consisting of spermicide and condom or diaphragm; using double-barrier contraception, specifically, a condom plus spermicide and a female diaphragm or cervical cap; using an approved intrauterine device (IUD) with established efficacy.
     3. Men, unless surgically sterilized (vasectomy with documentation of azoospermia), must agree to practicing abstinence or using barrier contraception, and not donate sperm, for a period of 6 months beginning from first dose of randomized treatment.

EXCLUSION CRITERIA:

1. General:

   1. Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
   2. Employees of Bristol-Meyers Squibb (BMS) or immediate family of BMS employees.
   3. Subjects with current participation in another clinical study in which the subject is or will be exposed to an investigational or non investigational drug or device; participation in a clinical study for an illness unrelated to alcohol use within the preceding month; or any previous participation in a trial involving pexacerfont or closely related compounds.
   4. Inability or unwillingness to participate in an MR scan, including presence of ferromagnetic metallic objects in the body, or pronounced claustrophobia
   5. Any medical or psychiatric condition or laboratory finding that, in the judgment of the investigator could adversely affect subject safety or study integrity.
   6. Subjects who are unlikely or unable to complete this study because of impending or likely incarceration while on the protocol.
   7. Subjects who are required to receive treatment by a court of law or involuntarily committed to treatment.
2. Sex and reproductive status:

   1. Inability or unwillingness to practice contraception as described above
   2. Women who are pregnant, breastfeeding, or planning to become pregnant within 6 months from the administration of first study drug dose.
   3. Men who are planning to father a child within 6 months from the

   administration of the first study drug dose
3. Exclusionary psychiatric conditions:

   1. Past or present diagnosis of schizophrenia, bipolar disease, or any psychotic disorder other than one determined to be substance induced; past or present diagnosis of dementia, or any other disorder which has led to a clinically significant cognitive impairment; any other psychiatric condition which at the present time requires, or in the past month has required pharmacological intervention other than standard withdrawal treatment as described in the NIAAA Assessment and Treatment Protocol (#05-AA-0121).
   2. A personality disorder which, in the investigator s judgment could lead to non-compliance with study procedures.
   3. Subjects, who in the investigator's judgment, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior in the last 6 months and/or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the last 2 months.
   4. Positive urine test for illegal drug use.
4. Exclusionary medical history and concurrent medical conditions:

   1. Subjects with clinically significant thyroid pathology that would interfere with efficacy or safety evaluations, or who are undergoing treatment for their thyroid pathology (e.g., thyroid supplementation).
   2. Subjects with adrenal or pituitary pathology as evidenced by medical history or suggested from abnormal screening laboratory tests.
   3. Subjects with a significant history (as judged by the Investigator) of seizure disorder (e.g., epilepsy or withdrawal seizures), other significant neurological disorders (e.g., Parkinson s Disease, multiple sclerosis, stroke, neurodegenerative disease, cerebral palsy) or severe head trauma.
   4. Subjects with active liver disease or a history of hepatic intolerance to medications that in the Investigator s judgment, is medically significant.
   5. Subjects with a history of Diabetes Mellitus Type I and II or gastric bypass or reduction surgery.
   6. Subjects with Human Immunodeficiency Virus (HIV) infection.
   7. Subjects with difficulty swallowing tablets or capsules.
5. Exclusionary physical and laboratory test findings

   1. QTc > 475 msec
   2. Platelets less than or equal to 75,000/mm(3)
   3. Hemoglobin less than or equal to 9g/dL
   4. Neutrophils, Absolute less than or equal to 1000/mm(3)
   5. SGOT (AST) > 3.0 times Upper Limit of Normal
   6. SGPT (ALT) > 3.0 times Upper Limit of Normal
   7. Bilirubin 2 times Upper Limit of Normal
   8. Creatinine greater than or equal to 2mg/dL
   9. Diastolic blood pressure > 105 mmHg
   10. TSH > 1.6 times Upper Limit of Normal
   11. Creatine kinase > 5 times Upper Limit of Normal
6. Prohibited treatments

   1. Regular use of psychotropic medication (antidepressant, lithium,

      antipsychotic, anxiolytic, antiepileptic, opiates, or hypnotics), within one week prior to inclusion, with the exception of benzodiazepines

      administered within the NIAAA program as part of alcohol withdrawal

      treatment. Fluoxetine may not have been taken within 5 weeks, and depot antipsychotics may not have been taken within 12 weeks.
   2. Any change in a non-excluded medication in the past 3 months.
   3. Systemic intake of corticosteroids acutely within two weeks or chronically within the last 6 months (Topical hydrocortisone and inhaled corticosteroids are allowed).
   4. Patients taking medications that are CYP3A4 inhibitors or inducers, should not be taking these medications for at least seven days prior to randomization and during the remainder of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Heilig, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Heilig M, Egli M. Pharmacological treatment of alcohol dependence: target symptoms and target mechanisms. Pharmacol Ther. 2006 Sep;111(3):855-76. doi: 10.1016/j.pharmthera.2006.02.001. Epub 2006 Mar 20. PMID 16545872
- [Background] Epstein DH, Preston KL, Stewart J, Shaham Y. Toward a model of drug relapse: an assessment of the validity of the reinstatement procedure. Psychopharmacology (Berl). 2006 Nov;189(1):1-16. doi: 10.1007/s00213-006-0529-6. Epub 2006 Sep 22. PMID 17019567
- [Background] Anton RF, Moak DH, Latham PK. The obsessive compulsive drinking scale: A new method of assessing outcome in alcoholism treatment studies. Arch Gen Psychiatry. 1996 Mar;53(3):225-31. doi: 10.1001/archpsyc.1996.01830030047008. PMID 8611059
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-AA-0010.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pexacerfont | Placebo
Started | 40 | 30
Scripts Challenge Sessions | 26 | 25
Measure Drug Level Concentration | 10 | 0 (No placebo subjects completed this milestone which measured active drug levels)
Completed | 38 (Two subjects did not complete the scripts sessions but completed the remainder of the protocol) | 25
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pexacerfont | Placebo | Total
Number analyzed (Participants) | 40 | 30 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 30 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 34 | 25 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 38 | 30 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 19 | 39
  White | 16 | 9 | 25
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: Alcohol craving was measured using the Alcohol Urges Questionnaire (AUQ). The AUQ is an 8-item self-administered instrument that assesses craving for alcohol among alcohol users in the current context (i.e., right now). The score ranges from 8 (lowest craving value) to 56 (highest craving value).
Time Frame: 15 minutes prior to the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
Units on a scale | 12.7 (2.48) | 10.7 (2.60)

2. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 18.7 (2.48) | 14.5 (2.6)

3. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
Units on a scale | 16.6 (2.48) | 12.9 (2.6)

4. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 16.5 (2.48) | 11.8 (2.6)

5. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 15 (2.48) | 12.1 (2.6)

6. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 13.7 (2.48) | 12.3 (2.6)

7. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 13.5 (2.48) | 12 (2.6)

8. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 13.7 (2.48) | 11.7 (2.6)

9. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes prior to the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 12.9 (2.61) | 10.2 (2.74)

10. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 17.8 (2.61) | 14.4 (2.74)

11. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 16.8 (2.61) | 12.5 (2.74)

12. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 15.3 (2.61) | 12.2 (2.74)

13. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 14.9 (2.61) | 11.6 (2.74)

14. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 14.3 (2.61) | 11.6 (2.74)

15. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 14.9 (2.61) | 11.7 (2.74)

16. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of script presentation, which occurred on Day 24, 25, or 26 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pexacerfont | Placebo
Number analyzed (Participants) | 26 | 25
Units on a scale | 14.6 (2.61) | 11.2 (2.74)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected biweekly throughout the 27 day inpatient stay, and at two follow-up outpatient visits at 1 and 4 weeks following discharge
Arm/Group | Pexacerfont | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/30
Other Adverse Events (participants affected / at risk) | 34/40 | 28/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pexacerfont (N=40) | Placebo (N=30)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 11
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 29 | 24
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 7 | 6
Headache (Nervous system disorders) | 23 | 23
Memory impairment (Nervous system disorders) | 0 | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No